CLINICAL TRIAL: NCT07086599
Title: Typological Study of Sleep Pathologies During Psoriatic Rheumatism and SAPHO Syndrome: Prospective Study Within the Paris Saint-Joseph Hospital Group"
Acronym: SleepSO2
Status: Recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 642-SleepSO2; 2023-A01037-38 (Other: ID RCB)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis Arthritis; SAPHO Syndrome; Sleep Apnea Syndromes
MeSH Terms: conditions — Acquired Hyperostosis Syndrome; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No sleep disorder
- sleep apnea
- other sleep disorder

SUMMARY:
Chronic inflammatory rheumatisms (CIR) are a source of motor disability and various comorbidities, particularly cardiovascular and metabolic. They also significantly impact patients' quality of life, including sleep disturbances. Among CIRs, psoriatic arthritis is a chronic inflammatory arthropathy associated with psoriasis, typically seronegative for rheumatoid factor. This heterogeneous disease affects peripheral and/or axial joints and can include extra-articular manifestations such as uveitis and chronic inflammatory bowel diseases. Its prevalence is estimated between 0.3% and 1% in the general population.

SAPHO syndrome, similar to psoriatic arthritis, is characterized by specific bone involvement with a hypertrophic tendency, often affecting the axial skeleton and the anterior thoracic wall. Pain and inflammation are closely linked to sleep quality, creating a vicious cycle where pain disrupts sleep and poor sleep amplifies pain perception. Analgesic treatments, such as opioids, can also cause nocturnal respiratory pathologies, further disrupting sleep.

Inflammatory processes are regulated by sleep, influencing plasma concentrations of CRP, IL6, and TNF production. Patients with psoriatic arthritis or SAPHO syndrome share common risk factors with Obstructive Sleep Apnea Syndrome (OSAS), such as obesity, hypertension, and metabolic syndrome.

Sleep disorders are common in the general population and likely underdiagnosed in these patients. Several studies suggest a link between sleep disorders and these rheumatic conditions, affecting quality of life and exacerbating symptoms. Questionnaires like the Epworth and Pichot scales provide a more precise evaluation of these symptoms. However, objective sleep exploration through polysomnography has never been conducted in these patients.

In summary, CIRs, particularly psoriatic arthritis and SAPHO syndrome, significantly impact patients' quality of life and sleep, necessitating appropriate evaluation and management of associated sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient diagnosed with psoriatic arthritis or SAPHO syndrome and followed at Paris Saint-Joseph Hospital
* Patient presenting sleep disorders warranting hospitalization for further -investigation of these disorders
* French-speaking patient
* Patient who does not oppose participation in the research protocol

Exclusion Criteria:

* Patient already followed for a sleep disorder
* Patient who underwent polysomnography in the last 2 years
* End-of-life patient
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient diagnosed with psoriasis arthritis or SAPHO syndrome and presenting sleep disorder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2027-05-13 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Type of sleep disorders | at 6months
  sleep disorders will be defined after polysomnography exam.

SECONDARY OUTCOMES:
sleep structure | at 6 months
  quantity of the different sleep stages as observed on the polysomnography exam
presence and severity of asthenia, | at enrollement
  mesured by the PICHOT questionnar
evaluation of anxiety | at enrollement
  mesured by HAD questionnaire
drowsiness evaluation | at enrollement
  mesured with the Epworth Scale
Evaluation of Sleep Apnea | at enrollement, at 6months and at 12 months
  mesured with the STOP BANG questionnaire
Sleep apnea severy | at enrollemnt, 6months and 12 months after
  mesured by the Apnea/hypopnea index
Rheumatism disease activity | at enrollement, after 6 months and after 12 months
  mesured with the DPASA score
CRP mesurement | at enrollment, 6months and 12 months after
  expressed in mg/L

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Paris Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No